CLINICAL TRIAL: NCT07079059
Title: Comparative Analysis of Virtual Reality Simulation Training on Clerkship Anesthesia Rotation Experience for Medical Students in a Canadian Setting
Brief Title: VR in Undergraduate Anesthesia Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Aldo Espinosa Tadeo, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VR in Anesthesia UGME
Record Dates: First submitted 2025-07-09; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia
Keywords: Virtual Reality; Undergraduate Medical Education; Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Training (Experimental): Students will complete a one-hour VR training session on the first day of their anesthesia rotation. Virtual reality-based training will use a high-fidelity VR simulation platform on Quest VR headsets, allowing students to practice key anesthesia skills, including airway management techniques (e.g., supraglottic airway placement, endotracheal intubation), anesthetic agent preparation and administration, and patient monitoring during anesthesia. questions. After completing the VR training, students will proceed with their standard two-week anesthesia rotation in clinical settings.
  Interventions: Other: Virtual Reality Training
- Standard Training (No Intervention): Students in this group will not receive VR training and will follow the existing standard teaching curriculum without any modification, which includes traditional didactic lectures and hands-on learning in the clinical setting under faculty supervision. All aspects of the student's training will remain the same and not be impacted by participation in this study.

INTERVENTIONS:
Other: Virtual Reality Training — One hour of virtual reality training to be included in students' Anesthesia training prior to the start of their Anesthesia rotation.
  Arms: Virtual Reality Training

SUMMARY:
Medical students learning anesthesia often face challenges in gaining hands-on experience due to the complexity of the operating room environment. Traditional teaching methods, such as lectures and in-person training, can be inconsistent due to variations in clinical exposure and instructor availability. Virtual reality (VR) technology offers an innovative solution by allowing students to practice anesthesia-related skills in a risk-free, immersive environment. This study will evaluate whether VR simulation training can better prepare third-year medical students for their anesthesia rotation compared to traditional methods. Students will be randomly assigned to one of two groups: one will receive VR training before their rotation, while the other will follow the standard curriculum without VR. To assess the effectiveness of VR training, all students will complete pre- and post-rotation surveys measuring their confidence in anesthesia principles, procedural skills, and overall preparedness. Additionally, faculty will use a standardized checklist to evaluate students' performance on key anesthesia procedures during their clinical rotations. By comparing students who received VR training to those who did not, this study will determine if VR can improve knowledge retention, skill development, and confidence in real clinical settings. If successful, VR technology could enhance anesthesia education and provide new training opportunities for medical students, including those in remote or resource-limited settings.

DETAILED DESCRIPTION:
Anesthesia rotations are complex and challenging, often intimidating for students due to their safety-critical environment. Traditional anesthesia teaching methods for medical students in Canada comes with several challenges such as variability in exposure for students, patient safety concerns with staff, and instructor availability. High-fidelity VR simulations provide an innovative, consistent, and engaging educational experience, allowing students to practice critical skills in a risk-free setting. The purpose of this study is to determine whether VR simulation training improves third-year medical students' perceptions on their clinical performance, confidence, and knowledge retention during anesthesia rotations compared to our current teaching methods. We hypothesize that VR training will result in superior outcomes in student performance and confidence during their Anesthesia rotation. The study will include 180 third-year medical students, randomly assigned to control and experimental groups.

This study involves third-year medical students as participants and will assess the impact of virtual reality (VR) simulation training on their confidence and preparedness for anesthesia rotations. After consent is obtained, participants will be randomly assigned to one of two groups:

1. Experimental Group (VR Training Group) Students will complete a one-hour VR training session on the first day of their anesthesia rotation. Prior to VR training, students in the VR training group will be asked to complete a short survey that will assess the participant's knowledge, confidence, and procedural skills as applicable to their upcoming Anesthesia rotation. This survey will take approximately 5-10 minutes to complete. Virtual reality-based training will use a high-fidelity VR simulation platform on Quest VR headsets, allowing students to practice key anesthesia skills, including airway management techniques (e.g., supraglottic airway placement, endotracheal intubation), anesthetic agent preparation and administration, and patient monitoring during anesthesia.

   A faculty member or research assistant will be available during the session to guide students and answer questions. After completing the VR training, students will proceed with their standard two-week anesthesia rotation in clinical settings. All other aspects of the student's training will remain the same and not be impacted by participation in this study.

   Following completion of the Anesthesia training rotation, participants will be asked to complete a post-rotation online survey. The post-rotation survey will assess knowledge, confidence, and procedural skills through self-rated confidence in anesthesia principles, pharmacology, monitoring, procedural skills (e.g., intubation, airway management and overall preparedness for the operating room. This survey will take approximately 5-10 minutes to complete.

   The VR device will be cleaned using disinfectant wipes between uses.
2. Control Group (Standard Training Group) Students in this group will not receive VR training and will follow the existing standard teaching curriculum without any modification, which includes traditional didactic lectures and hands-on learning in the clinical setting under faculty supervision. All aspects of the student's training will remain the same and not be impacted by participation in this study. Prior to commencing their anesthesia rotation, students will be asked to complete a short survey on that will assess their knowledge, confidence, and procedural skills as applicable to their upcoming Anesthesia rotation. This survey will take approximately 5-10 minutes to complete.

Participants will be asked to complete a post-rotation online survey. The post-rotation survey will assess knowledge, confidence, and procedural skills through self-rated confidence in anesthesia principles, pharmacology, monitoring, procedural skills (e.g., intubation, airway management and overall preparedness for the operating room. This survey will take approximately 5-10 minutes to complete.

Both groups will receive the same pre and post-rotation surveys to complete. The post-rotation survey will assess knowledge, confidence, and procedural skills through self-rated confidence in anesthesia principles, pharmacology, monitoring, procedural skills (e.g., intubation, airway management and overall preparedness for the operating room. The only difference will be that the VR simulation training group participants will indicate "yes" when asked if they underwent VR training which will trigger additional questions regarding their use of VR.

Both groups will also have data related to standard faculty assessments of their rotation performance collected to determine whether VR training had any impact on the participant's performance during their Anesthesia rotation. in addition, faculty will complete questions related to research-specific assessments of students that rate perceived confidence, procedural skills, and overall preparedness of students and will indicate whether they were aware of the student's training modality (VR or traditional) to account for potential bias. Open-ended questions will explore faculty perceptions of differences, improvements, or challenges related to VR-trained students. Ideally, faculty will be blinded to the training method to minimize bias. However, given the practical aspects of clinical teaching, blinding may not always be possible. Faculty will be asked whether they were aware of the student's VR training status. Faculty surveys will be administered after the rotation is complete to allow for a comprehensive assessment of student performance.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a third-year medical student in the Undergraduate Medical Education (UME) program at Western University (Schulich School of Medicine & Dentistry).
* Scheduled to complete a two-week anesthesia rotation at one of the affiliated teaching hospitals:

  * London: Victoria Hospital, St. Joseph's Hospital, or University Hospital
  * Windsor: Metropolitan Campus or Ouellette Campus
* Willing to participate in the study and provide informed consent.
* Able to complete pre- and post-rotation assessments (self-assessment surveys and procedural skills checklist) administered in the English language.
* 18 years of age or older

Exclusion Criteria:

* Prior clinical anesthesia experience before their core anesthesia rotation, including: Participation in an Optional Clinical Learning Opportunity (OCLO) in anesthesia. Completion of a summer elective or placement in anesthesia. Completion of an anesthesia selective before their core anesthesia rotation.
* Previous exposure to the VR training platform used in the study (e.g., prior experience with the specific VR simulation software for anesthesia training).
* Students who do not consent to participate in the study or do not wish to be randomized into either the VR or control group.
* Students unable to complete the study assessments in the English language, including: Pre- and post-rotation surveys. Observer-completed procedural skills checklist (during clinical rotations).
* Medical or personal conditions preventing participation, such as: severe motion sickness or vertigo that would prevent the use of VR headsets. Any condition that significantly impacts vision or motor function, affecting the ability to engage with VR simulations.
* Students who are experience nausea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Impact of virtual reality (VR) simulation on the confidence, preparedness, and procedural skill performance of third-year medical students during their anesthesia rotation. | Period of 2 weeks during the students' Anesthesia rotation
  This will be measured by analyzing student survey responses that self-report their perception of their confidence and preparedness in Anesthesia and their procedural skill performance as evaluated by Anesthesia Faculty preceptors.

SECONDARY OUTCOMES:
Perceived realism and usefulness of VR training | Period of 2 weeks during the students' Anesthesia rotation
  This will be measured by analyzing the data from post-rotation student surveys that will assess how realistic students found VR training compared to real-life scenarios and how useful students found VR training to be to prepare them for the Anesthesia rotation.
Feasibility of integrating VR into medical education | Period of 2 weeks during the students' Anesthesia rotation
  This will be measured by tracking drop-out rates to assess feasibility.
Identify factors that may influence training effectiveness | Period of 2 weeks during the students' Anesthesia rotation
  This will be measured by performing a sub-group analysis based on prior Anesthesia exposure, campus location, or learning preferences, as well as examining potential differences in outcomes (confidence, skill performance) based on these factors.
Barriers of integrating VR into medical education | Period of 2 weeks during the students' Anesthesia rotation
  This will be measured by analyzing the data from post-rotation student surveys that will assess student feedback on any potential barriers to adopting VR training in this setting.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Espinosa, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pottle J. Virtual reality and the transformation of medical education. Future Healthc J. 2019 Oct;6(3):181-185. doi: 10.7861/fhj.2019-0036. PMID 31660522
- [Background] Gu Y, Tenenbein M, Korz L, Busse JW, Chiu M. Simulation-based medical education in Canadian anesthesiology academic institutions: a national survey. Can J Anaesth. 2024 Dec;71(12):1725-1734. doi: 10.1007/s12630-024-02720-6. Epub 2024 Mar 7. PMID 38453798
- [Background] Duffy CC, Bass GA, Yi W, Rouhi A, Kaplan LJ, O'Sullivan E. Teaching Airway Management Using Virtual Reality: A Scoping Review. Anesth Analg. 2024 Apr 1;138(4):782-793. doi: 10.1213/ANE.0000000000006611. Epub 2023 Jul 19. PMID 37467164
- [Background] Jiang H, Vimalesvaran S, Wang JK, Lim KB, Mogali SR, Car LT. Virtual Reality in Medical Students' Education: Scoping Review. JMIR Med Educ. 2022 Feb 2;8(1):e34860. doi: 10.2196/34860. PMID 35107421
- [Background] Zheng T, Xie H, Gao F, Gong C, Lin W, Ye P, Liu Y, He B, Zheng X. Research and application of a teaching platform for combined spinal-epidural anesthesia based on virtual reality and haptic feedback technology. BMC Med Educ. 2023 Oct 25;23(1):794. doi: 10.1186/s12909-023-04758-4. PMID 37880665
- [Background] Palter VN, Grantcharov TP. Individualized deliberate practice on a virtual reality simulator improves technical performance of surgical novices in the operating room: a randomized controlled trial. Ann Surg. 2014 Mar;259(3):443-8. doi: 10.1097/SLA.0000000000000254. PMID 24503910
- [Background] Gan W, Mok TN, Chen J, She G, Zha Z, Wang H, Li H, Li J, Zheng X. Researching the application of virtual reality in medical education: one-year follow-up of a randomized trial. BMC Med Educ. 2023 Jan 3;23(1):3. doi: 10.1186/s12909-022-03992-6. PMID 36597093